CLINICAL TRIAL: NCT04360759
Title: Multi-centre Randomised Controlled Trial of Chloroquine/Hydroxychloroquine Versus Standard of Care for Treatment of Mild Covid-19 in HIV-positive Outpatients in South Africa
Brief Title: Chloroquine Outpatient Treatment Evaluation for HIV-Covid-19
Acronym: CQOTE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Equipoise for hydroxychloquine was lost
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Sean Wasserman, Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIV-COVID-19 CQOTE
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Covid-19; HIV
MeSH Terms: conditions — COVID-19 | interventions — Chloroquine; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Pragmatic, multi-centre, open label, randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Chloroquine or hydroxychloroquine (Experimental): Loading dose of 4 tablets (150 mg chloroquine base per chloroquine salt tablet; 155 mg chloroquine base per hydroxychloroquine tablet) at time 0 and 6 hours, followed by a maintenance dose of 2 tablets at time 12 hours, and then twice daily for a total of 7 days.
  Interventions: Drug: Chloroquine or hydroxychloroquine
- Arm 2: Standard of care (No Intervention): This does not include specific therapy under current guidelines.

INTERVENTIONS:
Drug: Chloroquine or hydroxychloroquine — Chloroquine has in vitro antiviral activity against many viruses, including SARS-CoV-1 and SARS-CoV-2. Chloroquine inhibits coronavirus replication at in vitro concentrations that are not cytotoxic and within a range of blood concentrations achievable during standard antimalarial treatment. Chloroquine inhibits viral replication through interference with glycosylation of coronavirus ACE2 receptors, required for viral entry, and downstream phagolysosome alkalisation, interfering with the low-pH-dependent steps of viral fusion and uncoating. Chloroquine also has anti-inflammatory properties and could provide benefit through this mechanism in Covid-19, where a cytokine storm has been described in critically ill patients. Hydroxychloroquine is a less toxic metabolite of chloroquine, has similar anti-inflammatory properties, and is more potent against SARS-CoV-2 in vitro.
  Arms: Arm 1: Chloroquine or hydroxychloroquine

SUMMARY:
Clinical manifestations of Covid-19 are poorly characterised in HIV co-infection, which may predispose to more severe disease. Reducing hospitalisation and severe illness in this population has important individual and public health benefits. The investigators propose a pragmatic multi-centre, randomized controlled trial in South Africa to evaluate the efficacy and safety of chloroquine or hydroxychloroquine to prevent progression of disease and hospitalisation amongst HIV-positive people with Covid-19 not requiring hospitalisation at initial assessment.

DETAILED DESCRIPTION:
The trial objective is to compare chloroquine (or hydroxychloroquine) versus standard of care for the primary endpoint of hospitalisation or death at 28 days. Consenting adults who meet criteria for a Covid-19 person under investigation and who are ≥18 years, known to be HIV-positive, not requiring immediate hospitalisation and are not at risk of cardiac toxicities related to the study drug will be enrolled. The total sample size will be 560 participants (280 in each arm).

ELIGIBILITY:
Inclusion Criteria:

* Tested for Covid-19 at a trial recruitment site as an outpatient;
* Age 18 years or older;
* Not requiring immediate hospitalisation;
* Mild disease, defined as respiratory rate <25/min, pulse rate <120/min, SpO2 >94%;
* HIV-positive by rapid test or documented history;
* Suspected or confirmed Covid-19;
* Signed informed consent.

Exclusion Criteria:

* Covid-19 diagnosed > 5 days prior to randomization;
* Active tuberculosis;
* Need for concomitant drugs that are contraindicated with the use of Chloroquine/hydroxychloroquine;
* QTcF interval > 480 ms;
* Known glomerular filtration rate < 10 ml/min;
* Known with glucose-6-phosphate dehydrogenase deficiency (G6PD);
* Previous adverse drug reaction to investigational product;
* Concurrent involvement in other research or use of chloroquine, hydroxychloroquine or any other 4-aminoquinolone or another experimental investigational medicinal product that is likely to interfere with the study medication.

Note: Pregnancy and breastfeeding are not exclusions for entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival at 28 days post-randomization between experimental group and standard of care group | Day 28
  Events defined as Hospitalisation or Death

SECONDARY OUTCOMES:
Incidence of serious adverse events | Day 28
Incidence of adverse events of special interest related to investigational product at time of hospitalisation | Day 28
Premature discontinuation of treatment | Day 28
Time from treatment initiation to death, ARDS (PF/SF ratio < 300), or mechanical ventilation | Day 28
Proportion with moderate and severe ARDS | Day 28
Duration of hospitalisation and ICU stay in survivors | Day 28
Incidence of Covid-19 in household contacts | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Sean Wasserman, MBChB, Principal Investigator — CIDRI-Africa, University of Cape Town; Graeme Meintjes, PhD, Principal Investigator — CIDRI-Africa, University of Cape Town
Locations (2):
- South Africa (2):
  - Khayelitsha Hospital, Cape Town, Western Cape
  - Groote Schuur Hospital, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Data collected from this study may be made available to other international researchers and institutions who are working to control this Public Health Emergency, but in a fully anonymized way. No personal identifiers will be available anywhere in the data. Dates will either not be included or will be shifted by a random interval so as to not make it possible to trace any identity.
Supporting Information: Study Protocol
Time Frame: Recruitment period is planned for a maximum of 12 months, rate dependent on patient numbers. Additional sites will be opened after initial approvals.